CLINICAL TRIAL: NCT04722445
Title: Diagnostic Accuracy of Early ulTrasound Measurement of Quadriceps Thickness During Neuromuscular EleCTrical Stimulation for the Diagnosis of ICU-acquired Weakness : an Observational Study (DETECT)
Brief Title: Ultrasound Measurement of Quadriceps Shortening During Neuromuscular Electrical Stimulation in Critically Ill Patients
Acronym: DETECT
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01690-39
Record Dates: First submitted 2020-10-22; First posted 2021-01-25 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: ICU Acquired Weakness; Quadriceps Muscle Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Early ultrasound measurement of quadriceps shortening during neuromuscular electrical stimulation (NMES) — NMES will be applied to the quadriceps muscle to generate muscle contraction. Ultrasound measurement of the quadriceps thickness will be provided during contraction and rest, and the shortening of the quadriceps muscle will be measured. A second measurement using Shear-wave elastography measurement will also be undertaken. The measures will be undertaken at day 1 of neuromuscular blockers liberation (if any) as well as at day 3 and day 7 for the patients that will still be received mechanical ventilation at that time.

SUMMARY:
ICU-Aw is highly prevalent (50%) among critically ill patients. Its diagnosis is usually delayed as it requires patients' awakening and collaboration to provide accurate measurement.

This study aims to investigate the accuracy of an early ultrasound measurement of quadriceps shortening during neuromuscular electrical stimulation to diagnose future ICU-Aw in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for at least 24 hours

Exclusion Criteria:

* Decision to withhold life-sustaining treatment
* Pregnancy
* Degenerative neurological pathology with disabling muscle weakness
* Pace Maker
* Inability to communicate
* Chronic loss of autonomy described by the patient's family
* Guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted in ICU departement and mechanically ventilated for at least 24 hours without counterindications to provide NMES.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
ICU-Aw diagnosis | In the 24 hours following extubation
  Measured with the Medical Research Council score (scored 0 (minimum) to 60 (maximum); with a score < 48 meaning ICU-acquired weakness)

SECONDARY OUTCOMES:
Respiratory muscles strength | In the 30 minutes before extubation (during spontaneous breathing trial)
  Maximal Inspiratory Pressure and Maximal Expiratory Pressure
Cough capacity | In the 30 minutes before extubation (during spontaneous breathing trial)
  Peak Cough Flow
Extubation failure/success | Within 48 hours after extubation
  Reintubation or death

CONTACTS AND LOCATIONS:
Overall Officials: Yann Combret, PhD, PT, Principal Investigator — Groupe Hospitalier du Havre
Locations (1):
- Groupe Hospitalier du Havre, Montivilliers, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning after publication and ending 60 months following article publication.
Access Criteria: For individual participant data meta-analysis. Proposals should be directed to yann.combret@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Medrinal C, Combret Y, Hilfiker R, Prieur G, Aroichane N, Gravier FE, Bonnevie T, Contal O, Lamia B. ICU outcomes can be predicted by noninvasive muscle evaluation: a meta-analysis. Eur Respir J. 2020 Oct 1;56(4):1902482. doi: 10.1183/13993003.02482-2019. Print 2020 Oct. PMID 32366493